CLINICAL TRIAL: NCT01204606
Title: Arthroscopic Rotator Cuff Repair With Multimodal Analgesia(MMA): A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Arthroscopic Rotator Cuff Repair With Multimodal Analgesia(MMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM-10-02
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMA group (Experimental)
  Interventions: Procedure: Arthroscopic rotator cuff repair with intraoperative periarticular injection
- Control group (Placebo Comparator)
  Interventions: Procedure: Arthroscopic rotator cuff repair with non-injection of MMA drugs

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair with intraoperative periarticular injection — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4 or 5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repaired of rotator cuff tear was done with suture anchors.
  * Mixed MMA drugs(ropivacaine 300mg;40ml, morphine 10mg;1ml, cefotetan 1g; dilution to ropivacaine, epinephrine 0.3mg;0.3ml, total volume:41.3ml) and sodium hyaluronate 20mg;2ml were injected divisionally periarticular area; intra-articular(sodium hyaluronate 20ml;2ml + 10.3ml); posterior joint capsule(10ml); subacromial space and around suprascapular nerve(11ml); anterior capsule(10ml).
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  * Peripheral intravenous PCA(Patient Controlled Analgesia) was connected.
  Arms: MMA group
Procedure: Arthroscopic rotator cuff repair with non-injection of MMA drugs — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4 or 5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repaired of rotator cuff tear was done with suture anchors.
  * 43.3ml of saline was injected divisionally periarticular area; intra-articular(12.3ml); posterior joint capsule(10ml); subacromial space and around suprascapular nerve(11ml); anterior capsule(10ml).
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  * Peripheral intravenous PCA(Patient Controlled Analgesia) was connected.
  Arms: Control group

SUMMARY:
* The purpose of this study is to compare the efficacy of periarticular injections consisting of ropivacaine, morphine, epinephrine, cefotetan, and hyaluronic acid with the efficacy of periarticular injections consisting of the same amount of placebo(isotonic saline) during arthroscopic rotator cuff repair.
* Adding of multimodal analgesia(MMA) to conventional rotator cuff repair, it was expected that could reduce postoperative pain and narcotic consumption.

ELIGIBILITY:
Inclusion Criteria:

* rotator cuff tear
* arthroscopic surgery

Exclusion Criteria:

* age<45 or >85
* allergies to the drugs used in the study
* acute trauma history
* history of renal disease
* history of hepatic disease
* osteoarthritis or rheumatic arthritis
* systemic condition with chronic pain
* history of infection
* could not understand the questions
* rotator cuff tear treated by the open technique, by debridement only

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) for Pain | postoperative 5 hours

SECONDARY OUTCOMES:
Postoperative narcotic consumption | every 6 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Jo, M.D., Ph.D, Principal Investigator — Seoul Metropolitan Government Seoul National University Boramae Medical Center; Joint and Spine Center
Locations (1):
- Joint and Spine Center; SMG-SNU Boramae Medical Center, Seoul, South Korea